CLINICAL TRIAL: NCT05090722
Title: A Pilot Study to Evaluate PureWick for Nocturia
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator changing locations.
Sponsor: Northwell Health (Other)
Collaborators: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-05023603
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- The PureWick Urine Collection System (Experimental): The PureWick Urine Collection System is intended for non-invasive urine output management. It pulls urine through tubing that is connected to a collection canister for proper disposal. It is designed to be used by patients, caregivers, or healthcare professionals in both home environments and professional care facilities.
  Interventions: Device: PureWick System

INTERVENTIONS:
Device: PureWick System — The PureWick system consists of the external catheter, collection tubing, and collection canister with lid. It operates via a power cord that is plugged into the device outlet and the A/C power outlet.
  Other Names: PureWick Urine Collection System device; PWF030F

SUMMARY:
This is a single-center prospective pilot study of PureWick used as a management for nocturia and reduction of nighttime falls associated with going to the bathroom. Subjects are followed up to 3 months after the intervention. As a pilot study, it is expected that a 3-month follow-up will adequately capture urinary and sleep outcomes data and any adverse events related or unrelated to the study device.

DETAILED DESCRIPTION:
Nocturia is a highly prevalent condition among older adults, significantly affecting the quality of life as well as putting them at an increased risk of falls and fractures. In those 65 and older, accidental falls are identified as the leading cause of injury and death. The chance of falling increases from 30% to 50% with age greater than 85 years.

A study identified that in 1508 ambulatory men and women, nighttime urination of 2 times at night is associated with increased risk of falls (OR=1.84, 95% CI 1.05-3.22), with significantly higher risks when it increased to 3 or more times at night (OR=2.15, CI 95% -1.04-4.44). Incontinence management that reduces the need to get out of bed will lead to reduced risk of falls and unintentional injury fatalities.

The PureWick Urine Collection System is intended for non-invasive urine output management. It pulls urine through tubing that is connected to a collection canister for proper disposal. It is designed to be used by patients, caregivers, or healthcare professionals in both home environments and professional care facilities.

The PureWick System allows individuals to void while still in bed, demonstrating the potential to reduce the risks of falls associated with nighttime voids in men and women with nocturia. We hypothesize that this will also improve sleep quality and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 50 years or older.
* Experiences 2 or more voids per night as assessed on a 3-day bladder diary.

Exclusion Criteria:

* Compromised skin integrity in the perineal area (e.g., ulcers, open wounds, etc.).
* Neurological impairment or psychiatric disorder preventing proper understanding of consent.
* Unable to operate the PureWick system.
* Unable to complete required questionnaires and diaries.
* Investigator deems subject as unsuitable for enrollment.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients at 3 months who have a demonstrated 50% or greater reduction in the number of nocturia episodes/night | 3 months
  The proportion of patients at 3 months who have a demonstrated 50% or greater reduction in the number of nocturia episodes/night will be calculated via binomial proportions and an exact (Clopper-Pearson) 95% confidence interval will be computed to assess the precision of the obtained estimate.
Change in average number of nocturnal voids at baseline and at 3 months | At baseline and 3 months
  The paired t-test or Wilcoxon signed-rank test will be used, as appropriate, to compare the average number of nocturnal voids between baseline and at 3 months.
Change of scores on the N-QoL at baseline and at 3-months | At baseline and 3 months
  N-QoL (Nocturia quality of life) score is determined by the n-qol short form. The ICIQ-Nqol is a patient-completed questionnaire evaluating quality of life (QoL) in patients with nocturia for use in research and clinical practice across the world. The ICIQ-Nqol is the N-QoL adapted for use within the ICIQ structure and provides a detailed and robust measure to assess the impact of nocturia on quality of life with particular reference to the effects on patient' lives of Nocturia and can be used as an outcome measure to assess impact of different treatment modalities.
  0-52 overall score with greater values indicating increased impact on quality of life Bother scale not incorporated into overall score but indicate impact of symptoms overall for the patient.
  Similar analyses to paired t-test or Wilcoxon signed-rank test will be performed to compare scores on the N-QoL, an self-reported sleep quality between baseline and at 3-months.

SECONDARY OUTCOMES:
Change in the incidence of urinary tract infection (UTI) at baseline and 3 months | At baseline and 3 months
  McNemar's chi-square test will be used to compare the incidence of UTI between baseline and at 3 months.
Change in the incidence of pressure ulcers/skin breakdown at baseline and 3 months | At baseline and 3 months
  McNemar's chi-square test will be used to compare pressure ulcers/skin breakdown between baseline and at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Chughtai, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiarelli PE, Mackenzie LA, Osmotherly PG. Urinary incontinence is associated with an increase in falls: a systematic review. Aust J Physiother. 2009;55(2):89-95. doi: 10.1016/s0004-9514(09)70038-8. PMID 19463079
- [Background] Centers for Disease Control and Prevention, N.C.f.I.P.a.C. Web-based Injury Statistics Query and Reporting System (WISQARS). December 7, 2014].
- [Background] Medical Advisory Secretariat. Prevention of falls and fall-related injuries in community-dwelling seniors: an evidence-based analysis. Ont Health Technol Assess Ser. 2008;8(2):1-78. Epub 2008 Oct 1. PMID 23074507
- [Background] Hunter KF, Voaklander D, Hsu ZY, Moore KN. Lower urinary tract symptoms and falls risk among older women receiving home support: a prospective cohort study. BMC Geriatr. 2013 May 15;13:46. doi: 10.1186/1471-2318-13-46. PMID 23672343
- [Background] Beeson T, Davis C. Urinary Management With an External Female Collection Device. J Wound Ostomy Continence Nurs. 2018 Mar/Apr;45(2):187-189. doi: 10.1097/WON.0000000000000417. PMID 29394218